CLINICAL TRIAL: NCT02933918
Title: Safety of Intranasal Irrigation Probiotics in Healthy Volunteers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Probionase Therapies Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PROB001
Record Dates: First submitted 2016-10-06; First posted 2016-10-14 (Estimated); Last update posted 2023-11-18 (Actual); Status verified 2019-08

CONDITIONS: Sinusitis
Keywords: Probiotics; Nasal Irrigation; Healthy Volunteers
MeSH Terms: conditions — Sinusitis | interventions — Probiotics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Probiotics (Experimental)
  Interventions: Other: Probiotics

INTERVENTIONS:
Other: Probiotics — Safety of nasal irrigation with probiotics in healthy volunteers

SUMMARY:
Chronic rhinosinusitis (CRS) is one of the most common chronic diseases, affecting the quality of life of patients who suffer. Despite medical and surgical treatments available, there are a significant number of people suffering from CRS refractory to these standard treatments.

A preliminary clinical trial conducted at CHUM Hôtel-Dieu, has allowed us to evaluate the therapeutic potential of intranasal irrigation of probiotics in patients with CRS. This treatment administered twice daily for 14 days was well tolerated and resulted in improved chronic rhinosinusitis symptoms.

Prior to deployment on a larger scale, the safety of this therapy must be confirmed in a healthy population, free of sinus disease. Therefore, this study aims to assess the safety of the use of probiotic intranasal irrigation in healthy volunteers.

DETAILED DESCRIPTION:
If the participant (healthy volunteer) agrees to participate in the study, and after signing the information consent form, her/his participation in this project will consist to receive the experimental treatment of probiotics, to come to four (4) medical assessment visits at CHUM, over a period of time of four (4) weeks, and answer to one (1) phone call.

This study will include five (5) periods :

1. Determination of eligibility period (Day 0)
2. Saline irrigation period (Day 0 to Day 7)
3. Elimination of saline period (Day 8 to Day 14)
4. Probiotic treatment period (Day 15 to Day 21)
5. Telephone follow-up period (Day 22 to Day 28)

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 18 and older.
* Participant in general good health.
* Absence of nasal and ear signs or symptoms.

Exclusion Criteria:

* Participant suffering from acute rhinosinusitis, chronic rhinosinusitis, symptomatic allergic rhinitis, or other sinus disease.
* Participant with diseases of the middle ear causing impairment of the eardrum or middle ear, or have had surgery of the middle ear previously, except myringotomy with insertion tube.
* Primary or acquired immunodeficiencies documented.
* Antibiotic intake within 30 days before enrollment.
* Unable to do nasal rinse.
* Pregnant woman.
* Smell score from UPSIT-40 under normal smell threshold (<34).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2018-05-17 (Actual); Primary Completion 2019-12-30 (Actual); Study Completion 2019-12-30 (Actual)

PRIMARY OUTCOMES:
Change in sense of smell using the "University of Pennsylvania smell identification test (UPSIT-40)" | Change from baseline sense of smell at Day 7and Day 14
  A smell test will be conducted using "scratch and sniff fragrance strips" (UPSIT-40), where 40 odors are presented. The participant must choose one of four choices for each odor, even if she/he is unable to identify the smell.

SECONDARY OUTCOMES:
Change in sino-nasal symptomatology using questionnaire | Change from baseline sino-nasal symptomatology at Day 7, Day 14 and Day 21
  This questionnaire evaluates 5 items (nasal congestion, facial pain, headache, need to blow nose, post-nasal drip) on 0-3 scale (0= none; 1=mild; 2=moderate; 3= severe).
Change in Eustachian tube symptomatology using a questionnaire of Eustachian Tube Dysfunction (ETDQ-7) | Change from baseline Eustachian tube symptomatology at Day 7, Day 14 and Day 21
  Using a questionnaire of Eustachian Tube Dysfunction (ETDQ-7).
Change in ear examination | Change from baseline ear examination at Day 7 and Day 14
Change in anterior rhinoscopy | Change from baseline anterior rhinoscopy at Day 7 and Day 14

OTHER OUTCOMES:
Change in microbiome composition | Change from baseline microbiome composition at Day 7 and Day 14
  Evaluation of the difference in the percentage of the bacterial population before and after treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Martin Yvon Desrosiers, MD, Study Chair — Probionase Therapies Inc.
Locations (1):
- Centre Hospitalier de l'Université de Montréal, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No